CLINICAL TRIAL: NCT03795064
Title: Immediate Versus Early Endovenous Ablation In Venous Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Toni Pihlaja, Vascular Specialist, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 268/2018
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Venous Ulcer
Keywords: Venous Ulcer; Venous Insufficiency of Leg; Varicose Veins
MeSH Terms: conditions — Varicose Ulcer; Varicose Veins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Patients in this group will be treated with foam sclerotherapy immediately in the first visit to outpatient clinic (immediate intervention).
  Interventions: Procedure: Foam sclerotherapy; Procedure: Endothermal ablation
- Early Intervention (Active Comparator): Patients in this group will be treated with foam sclerotherapy in the following visit to outpatient clinic at four weeks (early intervention).
  Interventions: Procedure: Foam sclerotherapy; Procedure: Endothermal ablation

INTERVENTIONS:
Procedure: Foam sclerotherapy — Foam sclerotherapy is used to all patients for endovenous ablation of insufficient veins in subulcer plexus area.
Procedure: Endothermal ablation — Endothermal ablation is performed in early setting when truncal vein(s) anatomy is suitable.

SUMMARY:
The study is conducted to assess the effects of immediately started foam sclerotherapy in venous ulcer compared to early intervention.

DETAILED DESCRIPTION:
Recently EVRA study showed that early endovenous ablation (foam sclerotherapy and/or endothermal ablation) is beneficial for venous ulcer healing. This randomized controlled trial is conducted to assess the effects of immediate foam sclerotherapy in the first visit to vascular outpatient clinic (immediate intervention). Patients in control group will receive foam sclerotherapy at four weeks (early intervention). Endothermal ablation is performed in early setting in both groups when truncal vein anatomy is suitable. The primary outcome for this study is the reduction of venous ulcer area at four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Venous ulcer > 1 month
* Ulcer area > 1cm2
* Palpable distal pulses / Ankle-brachial index > 0,8 / Toe-brachial index > 70mmhg (at least one criteria must be met)

Exclusion Criteria:

* Leg ulcers other than venous etiology
* Pregnancy
* General contraindications for foam sclerotherapy
* Ulcers requiring operation theater revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Venous ulcer area | 0 to 180 days
  Venous ulcer area measured from calibrated digital photograph.

SECONDARY OUTCOMES:
Time to ulcer healing | 0 to 360 days
  Complete re-epithelialisation of ulcer area.
Total time of active venous ulcer | 0 to 360 days
  Time from when ulcer was first time noticed to complete re-epithelialisation of ulcer area.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Vascular Department, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pihlaja T, Ohtonen P, Romsi P, Pokela M. Sub-ulcer foam sclerotherapy in patients with venous ulceration: A randomized controlled trial. Phlebology. 2025 Jun;40(5):324-329. doi: 10.1177/02683555241304030. Epub 2024 Nov 27. PMID 39601296